CLINICAL TRIAL: NCT02543658
Title: The Curative Effect and Security of Neostigmine Treatment of Acute Pancreatitis Combined With Intra-abdominal Hypertension
Brief Title: Neostigmine Treatment of Acute Pancreatitis Combined With Intra-abdominal Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Lingyu Luo, Physician-in-charge, The First Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAHONCU
Record Dates: First submitted 2015-08-27; First posted 2015-09-07 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Acute Pancreatitis; Intra-abdominal Hypertension
Keywords: Acute Pancreatitis; Intra-abdominal hypertension; Abdominal compartment syndrome; Curative Effect; Security; Neostigmine
MeSH Terms: conditions — Pancreatitis; Intra-Abdominal Hypertension | interventions — Neostigmine; Conservative Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neostigmine (Experimental): Intramuscular injection of neostigmine on the basis of conventional conservative treatment
  Interventions: Drug: Neostigmine Methylsulfate 1 MG/ML; Combination Product: Conservative treatment
- Conservative treatment (Other): Intragastric administration of paraffin oil, 50ml,once every 8 hours；gastrointestinal decompression with nasogastric tube and rectal tub; lycerin enema promotes defecation; patients with ascites undergo percutaneous puncture drainage. Other conservative medical treatment recommended by the guidelines.
  Interventions: Combination Product: Conservative treatment

INTERVENTIONS:
Drug: Neostigmine Methylsulfate 1 MG/ML — The initial dose was 1mg, intramuscular injection(IM) once every 12 hours. If there is no defecation after 12 hours, the dose is increased to 1mg IM once every 8 hours; if there is no defecation after 24 hours, the dose is increased to 1mg IM once every 6 hours. If the abdominal pressure drops below 12mmhg, neostigmine will be stopped, otherwise it will be used continuously for 7 days.
  Other Names: Prostigmin
  Arms: Neostigmine
Combination Product: Conservative treatment — Intragastric administration of paraffin oil, 50ml,once every 8 hours；gastrointestinal decompression with nasogastric tube and rectal tub; lycerin enema promotes defecation; patients with ascites undergo percutaneous puncture drainage. Other conservative medical treatment recommended by the guidelines.
  Other Names: Non-surgical treatment

SUMMARY:
Acute pancreatitis(A) often complicated with Intra-abdominal Hypertension. After the onset of acute pancreatitis, capillary leakage causing ascites,upper gastrointestinal tract obstruction and paralytic ileus leading to an elevated IAP, severe IAH leads to ACS with high mortality. Neostigmine is an anti-cholinesterase drugs, can enhance intestinal peristalsis, promote flatus defecation. The aim of this study was to determine the effect of neostigmine on reducing abdominal pressure and clinical prognosis in patients with AP by promoting intestinal peristalsis and defecation.

DETAILED DESCRIPTION:
Acute pancreatitis(AP) runs a severe course in around 20% of patients and is associated with a mortality up to 30%. Intra-abdominal hypertension(IAH）is a common complication of severe acute pancreatitis(SAP). The inflammation of the pancreas starts a cascade of pancreatic and visceral edema, acute peripancreatic fluid collections, capillary leakage causing ascites, paralytic ileus, and gastric dilatation by upper gastrointestinal tract obstruction leading to an elevated intra-abdominal pressure (IAP). A sustained or repeated pathological elevation in IAP ≥12 mmHg is defined as IAH, it generally occurs often within the first week after onset of SAP. Persistent and serious IAH (IAP >20 mmHg ) often leads to new onset organ failure or acute worsening of existing organ failure, which is defined as ACS and associated with a mortality rate of 49%.

In the past practice, many patients with ACS undergo decompressive laparotomy, which obviously has a risk of complications. Therefore, numerous medical, nonmedical, and minimally invasive therapies have been introduced. Neostigmine is an anti-cholinesterase drugs, can enhance intestinal peristalsis, promote flatus defecation. World Society for Abdominal Compartment Syndrome (WSACS)guidelines,suggest that neostigmine be used for the treatment of established colonic ileus not responding to other simple measures and associated with IAH.However, no data exist on the effects of pharmacologic promotility therapy on IAP or outcomes among those with IAH/ACS. The aim of this study was to evaluate the efficacy of neostigmine on reducing IAP in AP patients with IAH.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 year ;
2. The diagnosis of acute pancreatitis according to the revised Atlanta classification.
3. IAH is defined as IAP ≥ 12 mmHg by the World Society of Abdominal;Compartment Syndrome (WSACS);
4. After 24 hours of conventional treatment(such as gastrointestinal decompression or percutaneous drainage of ascites), the IAP of AP patients with IAH was still ≥ 12 mmHg;
5. The onset time of acute pancreatitis was within 2 weeks;
6. Signed the informed consent.

Exclusion Criteria:

1. Previous history of laparotomy;
2. Mechanical ileus or abdominal hemorrhage were considered clinically;
3. Those who have contraindications to neostigmine: 1) Patients with angina; 2) myocardial infarction; 3) ventricular tachycardia; 4) bradycardia; 5) acute circulatory failure; 6) epilepsy; 7) bronchial asthma; 8) mechanical intestinal obstruction; 9) urinary tract infarction; 10) hyperthyroidism; 11) serious arrhythmia; 12) bladder operation; 13) intestinal fistula;
4. Allergic to neostigmine;
5. Pregnant or lactating patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nonghua Lv, MD, Study Chair — the Frist Affiliated Hospital of Nanchang University
Locations (1):
- Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Vidal MG, Ruiz Weisser J, Gonzalez F, Toro MA, Loudet C, Balasini C, Canales H, Reina R, Estenssoro E. Incidence and clinical effects of intra-abdominal hypertension in critically ill patients. Crit Care Med. 2008 Jun;36(6):1823-31. doi: 10.1097/CCM.0b013e31817c7a4d. PMID 18520642
- [Background] Kasi PM. The use of intravenous neostigmine in palliation of severe ileus. Case Rep Gastrointest Med. 2013;2013:796739. doi: 10.1155/2013/796739. Epub 2013 Feb 14. PMID 23476830
- [Background] Tracey KJ. The inflammatory reflex. Nature. 2002 Dec 19-26;420(6917):853-9. doi: 10.1038/nature01321. PMID 12490958
- [Background] Borovikova LV, Ivanova S, Zhang M, Yang H, Botchkina GI, Watkins LR, Wang H, Abumrad N, Eaton JW, Tracey KJ. Vagus nerve stimulation attenuates the systemic inflammatory response to endotoxin. Nature. 2000 May 25;405(6785):458-62. doi: 10.1038/35013070. PMID 10839541
- [Background] Schneider L, Jabrailova B, Soliman H, Hofer S, Strobel O, Hackert T, Buchler MW, Werner J. Pharmacological cholinergic stimulation as a therapeutic tool in experimental necrotizing pancreatitis. Pancreas. 2014 Jan;43(1):41-6. doi: 10.1097/MPA.0b013e3182a85c21. PMID 24212240
- [Background] Shaikh N, Kettern MA, Hanssens Y, Elshafie SS, Louon A. A rare and unsuspected complication of Clostridium difficile infection. Intensive Care Med. 2008 May;34(5):963-6. doi: 10.1007/s00134-007-0922-6. Epub 2007 Nov 20. PMID 18026931
- [Background] Kirkpatrick AW, Roberts DJ, De Waele J, Jaeschke R, Malbrain ML, De Keulenaer B, Duchesne J, Bjorck M, Leppaniemi A, Ejike JC, Sugrue M, Cheatham M, Ivatury R, Ball CG, Reintam Blaser A, Regli A, Balogh ZJ, D'Amours S, Debergh D, Kaplan M, Kimball E, Olvera C; Pediatric Guidelines Sub-Committee for the World Society of the Abdominal Compartment Syndrome. Intra-abdominal hypertension and the abdominal compartment syndrome: updated consensus definitions and clinical practice guidelines from the World Society of the Abdominal Compartment Syndrome. Intensive Care Med. 2013 Jul;39(7):1190-206. doi: 10.1007/s00134-013-2906-z. Epub 2013 May 15. PMID 23673399
- [Background] van Brunschot S, Schut AJ, Bouwense SA, Besselink MG, Bakker OJ, van Goor H, Hofker S, Gooszen HG, Boermeester MA, van Santvoort HC; Dutch Pancreatitis Study Group. Abdominal compartment syndrome in acute pancreatitis: a systematic review. Pancreas. 2014 Jul;43(5):665-74. doi: 10.1097/MPA.0000000000000108. PMID 24921201
- [Background] Trikudanathan G, Vege SS. Current concepts of the role of abdominal compartment syndrome in acute pancreatitis - an opportunity or merely an epiphenomenon. Pancreatology. 2014 Jul-Aug;14(4):238-43. doi: 10.1016/j.pan.2014.06.002. Epub 2014 Jun 17. PMID 25062870
- [Background] Ponec RJ, Saunders MD, Kimmey MB. Neostigmine for the treatment of acute colonic pseudo-obstruction. N Engl J Med. 1999 Jul 15;341(3):137-41. doi: 10.1056/NEJM199907153410301. PMID 10403850
- [Derived] He W, Chen P, Lei Y, Xia L, Liu P, Zhu Y, Zeng H, Wu Y, Ke H, Huang X, Cai W, Sun X, Huang W, Sutton R, Zhu Y, Lu N. Randomized controlled trial: neostigmine for intra-abdominal hypertension in acute pancreatitis. Crit Care. 2022 Mar 3;26(1):52. doi: 10.1186/s13054-022-03922-4. PMID 35241135

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Sept 1, 2015, and Aug 15, 2017, we measured intra-abdominal pressure on patients with acute pancreatitis and selected patients with intra-abdominal hypertension, in the Pancreatic Intensive Care Unit of the Department of Gastroenterology, the First Affiliated Hospital of Nanchang University.
Pre-assignment Details: Acute pancreatitis patients with intra-abdominal hypertension were first treated with conventional non-surgical therapy(such as: Enteral decompression with nasogastric and rectal tube,Glycerin enema, percutaneous drainage of ascites) for 24 hours. After 24 hours, the intra-abdominal pressure was still above 12 mmHg and they were randomized.
Groups:
- Neostigmine: Intramuscular injection of neostigmine
  Neostigmine Methylsulfate 1 MG/ML: The initial dose was 1mg intramuscular injection, q12h. If there is no defecation after 12 hours, the dose is increased to 1mg intramuscular injection, Q8H; if there is no defecation after 24 hours, the dose is increased to 1mg intramuscular injection, Q6 H. If the abdominal pressure drops below 12mmhg, stop using the drug, otherwise, it will be used for 7 days.
  Conservative treatment recommended by the guidelines, such as maintain the negative balance of fluid after the early recovery of fluid to stabilize the circulation, and to take appropriate sedative and analgesic treatment; negative pressure of the nasogastric tube attracts the contents of the stomach, and the glycerin is enema through the anus to promote defecation.Patients with ascites underwent percutaneous drainage.
- The Traditional Treatment: Conservative treatment recommended by the guidelines, such as maintain the negative balance of fluid after the early recovery of fluid to stabilize the circulation, and to take appropriate sedative and analgesic treatment; negative pressure of the nasogastric tube attracts the contents of the stomach, and the glycerin is enema through the anus to promote defecation.Patients with ascites underwent percutaneous drainage.
Period: Overall Study
Arm/Group | Neostigmine | The Traditional Treatment
Started | 40 | 40
Completed | 40 | 36
Not Completed | 0 | 4
Not completed — Lack of Efficacy | 0 | 4

BASELINE CHARACTERISTICS:
Population: A total of 80 out of 186 patients were included
Groups:
- Neostigmine: Intramuscular injection of neostigmine on the basis of conventional conservative treatment
  Neostigmine Methylsulfate 1 MG/ML: The initial dose was 1mg intramuscular injection, q12h. If there is no defecation after 12 hours, the dose is increased to 1mg intramuscular injection, Q8H; if there is no defecation after 24 hours, the dose is increased to 1mg intramuscular injection, Q6 H. If the abdominal pressure drops below 12mmhg, stop using the drug, otherwise, it will be used for 7 days.
  Conservative treatment: Intragastric administration of paraffin oil, 50ml, Q8H, gastrointestinal decompression with nasogastric tube and rectal tub; lycerin enema promotes defecation.; patients with ascites undergo percutaneous puncture drainage. Other conservative medical treatment recommended by the guidelines.
- Conservative Treatment: Intragastric administration of paraffin oil, 50ml, Q8H, gastrointestinal decompression with nasogastric tube and rectal tub; lycerin enema promotes defecation.; patients with ascites undergo percutaneous puncture drainage. Other conservative medical treatment recommended by the guidelines.
- Total: Total of all reporting groups
Arm/Group | Neostigmine | Conservative Treatment | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: yeas] | 46 (13) | 49 (14) | 48 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 27 | 34 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 40 | 40 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 40 | 40 | 80
Cause of pancreatitis [Count of Participants; unit: Participants]
  Biliary | 12 | 14 | 26
  Hyperlipidemic | 21 | 20 | 41
  Alcoholic | 4 | 4 | 8
  Idiopathic | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of IAP After Treatment
Description: Monitor the intra-abdominal pressure within 1 to 7 days after randomization, and calculate the percent change compared with that before randomization
Time Frame: From randomization to 7 days after treatment,Measured IAP every 6 hours
Population: The primary outcome measure was decreased rate of IAP after randomisation.
Measure: Median (Inter-Quartile Range); unit: percent change of IAP
Groups:
- Conservative Treatment: Intragastric administration of paraffin oil, 50ml, Q8H, gastrointestinal decompression with nasogastric tube and rectal tub; lycerin enema promotes defecation.; patients with ascites undergo percutaneous puncture drainage. Other conservative medical treatment recommended by the guidelines.
  Conservative treatment: Intragastric administration of paraffin oil, 50ml, Q8H, gastrointestinal decompression with nasogastric tube and rectal tub; lycerin enema promotes defecation.; patients with ascites undergo percutaneous puncture drainage. Other conservative medical treatment recommended by the guidelines.
Arm/Group | Neostigmine | Conservative Treatment
Number analyzed (Participants) | 40 | 40
percent change of IAP
  percent change of IAP at 24 hours | -18.7 [-28.4 to -4.7] | -5.4 [-18.0 to 0]
  percent change of IAP at 7 days | -27.2 [-39.4 to -5.3] | -20.0 [-26.7 to -5.9]

2. Secondary Outcome: The Change of Stool Volume at 1-7 Days After Randomization
Description: After randomization, the change of stool volume (ML) was calculated every 24 hours.For example, the amount of stool volume decreased or increased in 24 hours after grouping compared to before grouping.
Time Frame: From randomization to 7 days
Measure: Median (Inter-Quartile Range); unit: ml/day
Arm/Group | Neostigmine | Conservative Treatment
Number analyzed (Participants) | 40 | 40
ml/day
  The change of stool volume at 24 hours | 870 [250 to 2070] | 60 [-30 to 770]
  The change of stool volume at 7th day | 1025 [450 to 1520] | 370 [150 to 1200]

3. Secondary Outcome: New-onset Abdominal Compartment Syndrom
Description: Abdominal compartment syndrome is defined as a sustained IAP>20 mmHg (with or without an APP<60 mmHg) that is associated with new organ dysfunction/failure
Time Frame: From randomization to discharge or death, assessed up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Neostigmine | Conservative Treatment
Number analyzed (Participants) | 40 | 40
Participants | 2 | 4

4. Secondary Outcome: New-onset Organ Failure
Description: Incidence of organ failure from randomization to discharge or death, assessed up to 3 months
Time Frame: From randomization to discharge or death, assessed up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Neostigmine | Conservative Treatment
Number analyzed (Participants) | 40 | 40
Participants | 12 | 16

5. Secondary Outcome: Death of 90 Days
Description: Death during from randomization to 90 days after onset.
Time Frame: From randomization to 90 days after onset.
Measure: Count of Participants; unit: Participants
Arm/Group | Neostigmine | Conservative Treatment
Number analyzed (Participants) | 40 | 40
Participants | 10 | 11

6. Secondary Outcome: Timing of Enteral Nutrition
Description: From date of randomization to enteral nutrition, assessed up to 30 days
Time Frame: Start time of enteral nutrition after randomization, assessed up to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Neostigmine | Conservative Treatment
Number analyzed (Participants) | 40 | 40
days | 3 [3 to 4] | 4 [3 to 6]

7. Secondary Outcome: Number of Participants With Deterioration of IAH
Description: IAP rebound ≥ 5mmHg or increase ≥ 20mmHg within 1-7 days after grouping
Time Frame: From randomization to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Neostigmine | Conservative Treatment
Number analyzed (Participants) | 40 | 40
Participants | 4 | 8

8. Secondary Outcome: Number of Participants With Adverse Effects on the Cardiovascular System
Description: Due to that neostigmine has an inhibitory effect on the cardiovascular system, new-onset cardiovascular failure after grouping is considered as a possible adverse event related to neostigmine.Cardiovascular failure was defined as circulatory systolic blood pressure <90 mm Hg, despite adequate fluid resuscitation, or need for inotropic catecholamine support
Time Frame: From randomization to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Neostigmine | Conservative Treatment
Number analyzed (Participants) | 40 | 40
Participants | 8 | 4

9. Other Pre Specified Outcome: Days in Hospital
Description: Days in hospital within 6 months after randomisation
Time Frame: From randomisation to 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Neostigmine | Conservative Treatment
Number analyzed (Participants) | 40 | 40
days | 20 [13 to 31] | 19 [14 to 27]

10. Other Pre Specified Outcome: Days in ICU
Description: Days in ICU within 6 months after randomisation
Time Frame: From randomisation to 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Neostigmine | Conservative Treatment
Number analyzed (Participants) | 40 | 40
days | 12 [7 to 19] | 12 [8 to 15]

11. Other Pre Specified Outcome: Medical Expenses
Description: Medical expenses within 6 months after randomisation
Time Frame: From randomisation to 6 months
Measure: Median (Inter-Quartile Range); unit: thousand(RMB)
Arm/Group | Neostigmine | Conservative Treatment
Number analyzed (Participants) | 40 | 40
thousand(RMB) | 95.3 [58.7 to 146.8] | 102.3 [56.0 to 186.6]

ADVERSE EVENTS:
Time Frame: 6 months
Description: The main adverse events observed were the effects of neostigmine on the cardiovascular system, such as arrhythmias and decreased blood pressure
Arm/Group | Neostigmine | The Traditional Treatment
All-Cause Mortality (participants affected / at risk) | 10/40 | 11/40
Serious Adverse Events (participants affected / at risk) | 8/40 | 4/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neostigmine (N=40) | The Traditional Treatment (N=40)
Single cardiovascular failure (Cardiac disorders) | 3 (3) | 3 (3) — Emerging cardiovascular failure after randomization,
Cardiovascular and respiratory failure (Cardiac disorders) | 2 (2) | 0 (0) — Patient has both cardiovascular and respiratory failure
Cardiovascular and renal failure (Cardiac disorders) | 1 (1) | 1 (1) — The patient has both cardiovascular and renal failure
Cardiovascular, respiratory and renal failure (Cardiac disorders) | 2 (2) | 0 (0) — The patient has both cardiovascular, respiratory and renal failure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT02543658/Prot_SAP_000.pdf